CLINICAL TRIAL: NCT02974660
Title: Use of Protamine Sulfate During Transcatheter Aortic Valve Implantation - Impact on Bleeding and Thromboembolic Complications
Brief Title: Protamine Sulfate During Transcatheter Aortic Valve Implantation
Acronym: PS TAVI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WUM-KZ
Record Dates: First submitted 2016-10-10; First posted 2016-11-28 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Protamines; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protamine sulfate (Active Comparator): After obtaining optimal valve deployment patients will receive protamine sulfate (1 mg for each 100 units of UFH i.v.). Measurement of activated clotting time (ACT) will be performed (after heparin administration and after protamine sulfate administration).
  Interventions: Drug: Protamine sulfate
- 0.9% NaCl (Placebo Comparator): After obtaining optimal valve deployment patients will receive 0.9% saline (20 ml i.v.). Measurement of activated clotting time (ACT) will be performed (after heparin administration and after placebo administration).
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: Protamine sulfate
  Arms: Protamine sulfate
Drug: 0.9% NaCl
  Arms: 0.9% NaCl

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is a new, rapidly emerging standard of care in inoperable and high-risk patients with severe, symptomatic aortic stenosis. Information regarding reversal of unfractionated heparin with protamine sulfate in order to facilitate access site closure is scarce and based on expert consensus. Clinical practice varies between centers. Protamine sulphate may decrease the amount of bleeding complications related to the access-site. The impact on possible thromboembolic complications is unknown. Both bleeding and thromboembolic complications increase mortality after TAVI. A randomized trial is required in order to assess impact of protamine sulfate on prevalence and extent of bleeding and thromboembolic complications.

DETAILED DESCRIPTION:
Information regarding reversal of unfractionated heparin (UFH) with protamine sulfate (PS) is based on expert consensus from 2012, which recommends use of UFH in order to achieve activated clotting time (ACT) > 300 seconds as well as UFH reversal with PS in case of TAVI via transapical access as well as transfemoral access with the exception of cases with minimal bleeding risk. However, the clinical practice varies between centers - some use PS routinely, others - only in selected cases. The actual impact of PS on bleeding complications reduction is unknown. Furthermore, a pro-thromboembolic effect of the PS cannot be excluded. Both bleeding (major and life-threatening according to Valve Academic Research Consortium [VARC] criteria) and thromboembolic complications increase mortality after TAVI. The occurrence of these complications in international TAVI registries in 30-day observation ranges from 9.7% in case of major bleeding, 4.7% in case of life-threatening bleeds and 5% in case of strokes. There are no randomized studies assessing impact of PS on frequency of bleeding and thromboembolic complications after TAVI, its side-effects and influence on mortality. Randomized trial is required in order to assess impact of protamine sulfate on prevalence of bleeding and thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent successful TAVI
* with any approved TAVI device
* via transfemoral access
* with use of any of the approved vascular closure devices
* provided written informed consent

Exclusion Criteria:

* no consent
* periprocedural complications requiring continuation of heparin or administration of protamine sulfate
* alergy to fish, protamine, protamine derivates, history of Humulin N, Novolin N, Novolin NPH, Gensulin N, SciLin N, NPH Iletin II and isophane insulin intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12; Primary Completion 2020-07 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Bleeding complications | 48 hours or hospital discharge, whichever occurs first
  Composite of life-threatening and major bleeding complications according to Valve Academic Research Consortium (VARC) criteria (unit of measure: 0/1 [absence/presence])

SECONDARY OUTCOMES:
Successful closure of the access-site | 15 minutes
  Angiographic assessment of contrast extravasation from the access site after closure with preclose device at the end of the procedure. Unit of measure: 0/1 (absence/presence).
Thromboembolic complications | 5 days or hospital discharge, whichever occurs first
  Clinical assessment of thromboembolic complications in the central nervous system and peripheral vasculature (e.g. mesenteric, extremities). Unit of measure: 0/1 (absence/presence)
Assessment of peri-procedural myocardial muscle injury | 24 hours
  Measurements of levels of high sensitivity cardiac troponin T and isoenzyme MB of creatine kinase before the procedure and 6- and 12-24 hours after the procedure. Unit of measure: high sensitivity cardiac troponin T [ng/L], isoenzyme MB of creatine kinase [mcg/L].
All-cause mortality | 30 days
  All-cause mortality. Unit of measure: 0/1 (absence/presence).

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. Eur Heart J. 2012 Oct;33(19):2403-18. doi: 10.1093/eurheartj/ehs255. PMID 23026477
- [Result] Holmes DR Jr, Mack MJ, Kaul S, Agnihotri A, Alexander KP, Bailey SR, Calhoon JH, Carabello BA, Desai MY, Edwards FH, Francis GS, Gardner TJ, Kappetein AP, Linderbaum JA, Mukherjee C, Mukherjee D, Otto CM, Ruiz CE, Sacco RL, Smith D, Thomas JD, Harrington RA, Bhatt DL, Ferrari VA, Fisher JD, Garcia MJ, Gardner TJ, Gentile F, Gilson MF, Hernandez AF, Jacobs AK, Kaul S, Linderbaum JA, Moliterno DJ, Weitz HH; American Heart Association; American Society of Echocardiography; European Association for Cardio-Thoracic Surgery; Heart Failure Society of America; Mended Hearts; Society of Cardiovascular Anesthesiologists; Society of Cardiovascular Computed Tomography; Society for Cardiovascular Magnetic Resonance. 2012 ACCF/AATS/SCAI/STS expert consensus document on transcatheter aortic valve replacement: developed in collabration with the American Heart Association, American Society of Echocardiography, European Association for Cardio-Thoracic Surgery, Heart Failure Society of America, Mended Hearts, Society of Cardiovascular Anesthesiologists, Society of Cardiovascular Computed Tomography, and Society for Cardiovascular Magnetic Resonance. J Thorac Cardiovasc Surg. 2012 Sep;144(3):e29-84. doi: 10.1016/j.jtcvs.2012.03.001. No abstract available. PMID 22898522
- [Result] Rodes-Cabau J, Dauerman HL, Cohen MG, Mehran R, Small EM, Smyth SS, Costa MA, Mega JL, O'Donoghue ML, Ohman EM, Becker RC. Antithrombotic treatment in transcatheter aortic valve implantation: insights for cerebrovascular and bleeding events. J Am Coll Cardiol. 2013 Dec 24;62(25):2349-2359. doi: 10.1016/j.jacc.2013.03.029. Epub 2013 Apr 10. PMID 23583252
- [Result] Linke A, Wenaweser P, Gerckens U, Tamburino C, Bosmans J, Bleiziffer S, Blackman D, Schafer U, Muller R, Sievert H, Sondergaard L, Klugmann S, Hoffmann R, Tchetche D, Colombo A, Legrand VM, Bedogni F, lePrince P, Schuler G, Mazzitelli D, Eftychiou C, Frerker C, Boekstegers P, Windecker S, Mohr FW, Woitek F, Lange R, Bauernschmitt R, Brecker S; ADVANCE study Investigators. Treatment of aortic stenosis with a self-expanding transcatheter valve: the International Multi-centre ADVANCE Study. Eur Heart J. 2014 Oct 7;35(38):2672-84. doi: 10.1093/eurheartj/ehu162. Epub 2014 Mar 28. PMID 24682842
- [Result] Borz B, Durand E, Godin M, Tron C, Canville A, Litzler PY, Bessou JP, Cribier A, Eltchaninoff H. Incidence, predictors and impact of bleeding after transcatheter aortic valve implantation using the balloon-expandable Edwards prosthesis. Heart. 2013 Jun;99(12):860-5. doi: 10.1136/heartjnl-2012-303095. Epub 2012 Dec 12. PMID 23236027
- [Result] Gauthier C, Astarci P, Baele P, Matta A, Kahn D, Kefer J, Momeni M. Mid-term survival after transcatheter aortic valve implantation: Results with respect to the anesthetic management and to the access route (transfemoral versus transapical). Ann Card Anaesth. 2015 Jul-Sep;18(3):343-51. doi: 10.4103/0971-9784.159804. PMID 26139739
- [Derived] Zbronski K, Grodecki K, Gozdowska R, Ostrowska E, Wysinska J, Rymuza B, Scislo P, Wilimski R, Kochman J, Filipiak KJ, Opolski G, Huczek Z. Protamine sulfate during transcatheter aortic valve implantation (PS TAVI) - a single-center, single-blind, randomized placebo-controlled trial. Kardiol Pol. 2021;79(9):995-1002. doi: 10.33963/KP.a2021.0070. Epub 2021 Jul 22. PMID 34292562